CLINICAL TRIAL: NCT01554722
Title: Incidence of Intraneural Needle Insertion in Ultrasound Guided Femoral Block: Out of Plane Versus in Plane Approach
Brief Title: Needle Nerve Contact in Ultrasound Guided Femoral Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Ana Ruiz, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R6345
Record Dates: First submitted 2012-02-27; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Peripheral Nerve Injury
Keywords: Ultrasound guidance; Femoral nerve block; Needle placement; Intraneural needle insertion
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- in plane needle placement (Experimental)
  Interventions: Procedure: Needle placement
- out of plane needle placement (Experimental)
  Interventions: Procedure: Needle placement

INTERVENTIONS:
Procedure: Needle placement — In plane versus out of plane needle placement techniques

SUMMARY:
Ultrasound-guided femoral nerve block is a common regional anesthesia technique. The optimal method of needle guidance (in-plane versus out-of-plane) with regards to the block efficacy and avoidance of needle-nerve contact has not been established. In this study the investigators tests the hypothesis that the incidence of needle-nerve contact is higher with the needle insertion in an out-of-plane than with the in-plane approach.

DETAILED DESCRIPTION:
Fourty-four patients with hip fracture (American Society of Anesthesiologists physical status 1-3) are being randomized to receive the femoral block with an out-of-plane (needle inserted at a 45°-60° angle 1 cm caudal to the midpoint of the ultrasound probe just above the femoral nerve) or an in-plane technique (needle inserted 0.5 cm from the side of the probe lateral to the femoral nerve). The data collected includes the depth of needle insertion at the endpoint before injection, response to nerve stimulation, distribution of the injected volume in relation to the nerve (anterior vs posterior, the latter indicating impalement), block efficacy at 20 minutes and 24 hours, and any signs of nerve injury).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3 patients
* Diagnosis of trochanteric or cervical hip fracture
* Hip replacement under spinal anesthesia

Exclusion Criteria:

* Patients under the age of 65 years or over the age of 90 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Number of intraneural needle insertion in ultrasound-guided femoral block: out-of-plane versus in-plane approach | 4 months
  The incidence of needle-nerve contact is higher with the out-of-plane approach (inserting the needle into the fascia at the midpoint over the femoral nerve)needle-nerve contact than with the in-plane approach (inserting the needle lateral to the femoral nerve).

SECONDARY OUTCOMES:
Number of Participants with femoral block success in ultrasound-guided femoral block: out-of-plane versus in-plane approach. | 4 months
  The efficacy of the out-of-plane approach (inserting the needle into the fascia at the midpoint over the femoral nerve)needle-nerve contact and the in-plane approach (inserting the needle lateral to the femoral nerve).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Sala-Blanch, MD, Principal Investigator — University Clinic Barcelona; Ana Ruiz, MD, Principal Investigator — University of Barcelona; Julia Martinez-Ocon, MD, Study Chair — University of Barcelona; Maria J Carretero, MD, Study Chair — University of Barcelona; Gerard Sánchez-Etayo, MD, Study Chair — University of Barcelona; Admir Hadzic, Prof Dr, Study Director — Columbia University St Luke's Hospital
Locations (2):
- St Luke'S Roosevelt Hospital, Columbia University, New York, New York, United States
- University of Barcelona, Barcelona, Spain